CLINICAL TRIAL: NCT04191603
Title: THE EFFECTIVENESS OF MONOPOLAR HOOC VERSUS PLASMAKINETIC BİPOLAR SPATULA USAGE DURING COLPOTOMY PROCESS IN PATIENTS UNDERGOİNG TOTAL LAPAROSCOPIC HYSTERECTOMY
Brief Title: TWO DİFFERENT ELECTROSURGERY DEVICES AS MONOPOLAR HOOC AND PLASMAKINETIC BIPOLAR SPATULA EFFECTIVENESS DURING COLPOTOMY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alkü Alanya Education and Research Hospital (Other)
Responsible Party: Principal Investigator, MERAL TUĞBA ÇİMŞİR, ASSOCIATE PROFESSOR, Alkü Alanya Education and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: ALKU ERH
Record Dates: First submitted 2019-12-04; First posted 2019-12-10 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Uterine Fibroid; Ovary Cyst; Endometrial Hyperplasia; Cervical Dysplasia
MeSH Terms: conditions — Leiomyoma; Ovarian Cysts; Endometrial Hyperplasia; Uterine Cervical Dysplasia

STUDY DESIGN:
Intervention Model Description: MONOPOLAR HOOC VERSUS PLASMAKINETIC BIPOLAR SPATULA USAGE DURING COLPOTOMY
Who Masked: Investigator
Masking Description: MONOPOLAR HOOC VERSUS PLASMAKINETIC BIPOLAR SPATULA USAGE DURING COLPOTOMY
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MONOPOLAR HOOC (Active Comparator): COLPOTOMY WITH USAGE MONOPOLAR HOOC
  Interventions: Device: MONOPOLAR HOOC
- PLASMAKINETIK BIPOLAR SPATULA (Active Comparator): COLPOTOMY WITH USAGE MONOPOLAR HOOC
  Interventions: Device: PLASMAKINETIC BIPOLAR SPATULA

INTERVENTIONS:
Device: MONOPOLAR HOOC — COLPOTOMY WITH MONOPOLAR HOOC
  Arms: MONOPOLAR HOOC
Device: PLASMAKINETIC BIPOLAR SPATULA — COLPOTOMY WITH BIPOLAR SPATULA
  Arms: PLASMAKINETIK BIPOLAR SPATULA

SUMMARY:
WE DECIDED TO COMPARE TWO DIFFERENT ELECTROSURGERY DEVİCES TO PROVIDE COLPOTOMY. ONE OF THEM İS MONOPOLAR HOOC, THE OTHER DEVİCE İS PLASMAKİNETİC BİPOLAR SPATULA. WE WİLL RANDOMİSE PATİENTS FİRSTLY THEN COMPARE THE RESULTS SUCH, VAGİNAL DEHİSSENS, COLPOTOMY DURATİON, AMOUNT OF MIST DURING COLPOTOMY, AMOUNT OF BLEEDİNG.

DETAILED DESCRIPTION:
COLPOTOMY IS A PROCESS DURING TOTAL LAPAROSCOPIC HYSTERECTOMY. WE CAN USE EİTHER ELECTROSURGERY INSTRUMENTS TO PROVIDE COLPOTOMY. IN OUR TRIAL WE WİLL RANDOMİSE PATİENTS FİRSTLY THEN COMPARE THE RESULTS SUCH, VAGİNAL DEHİSSENS, COLPOTOMY DURATİON, AMOUNT OF MIST DURING COLPOTOMY, AMOUNT OF BLEEDİNG.

ELIGIBILITY:
Inclusion Criteria:

* APPROPIATE FOR TOTAL LAPAROSCOPIC HYSTERECTOMY

Exclusion Criteria:

* MALIGNANCY

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10-30 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
VAGINAL DEHISSENS | 0 DAY-365 DAYS
  AFTER LAPAROSCOPIC HYSTERECTOMY TWO DIFFERENT ELECTROSURGERY DEVICES RESULTS

CONTACTS AND LOCATIONS:
Overall Officials: MERAL TUĞBA ÇİMŞİR, Principal Investigator — ALKU EDUCATİON AND RESEARCH HOSPITAL
Locations (1):
- Alku Alanya Education and Research Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
5 YEARS
Supporting Information: CSR
Time Frame: 5 YEARS